CLINICAL TRIAL: NCT05897125
Title: TELE-TOC: Telehealth Education Leveraging Electronic Transitions Of Care for COPD Patients
Brief Title: Telehealth Education Leveraging Electronic Transitions Of Care for COPD Patients
Acronym: TELE-TOC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Washington University School of Medicine (Other); Society of Hospital Medicine (Other); COPD Foundation (Other); Hospital Medicine Reengineering Network (HOMERuN) (Unknown); The American Telemedicine Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB21-1325
Record Dates: First submitted 2023-05-10; First posted 2023-06-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: COPD Exacerbation; Care Transitions
Keywords: Medication education; Medication reconciliation; Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Investigator
Masking Description: Investigators will remain masked to treatment group and data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TELE-TOC plus Usual Care (Experimental): Patients randomized to this arm will receive the TELE-TOC intervention as well as the standard COPD care via the institution's COPD readmission reduction program.
  Interventions: Other: Virtual at Home Medication Reconciliation Visit(s); Behavioral: Virtual At Home Medication Education Visit(s); Other: COPD advanced practice nurse Inpatient Consult; Other: Inpatient Medication Reconciliation; Other: Post-discharge nurse 48 hour phone follow-up call; Other: Post-discharge follow-up advanced practice nurse outpatient visit
- Usual Care (Active Comparator): Patients randomized to this arm will receive standard COPD care via the institution's COPD readmission reduction program.
  Interventions: Other: COPD advanced practice nurse Inpatient Consult; Other: Inpatient Medication Reconciliation; Other: Post-discharge nurse 48 hour phone follow-up call; Other: Post-discharge follow-up advanced practice nurse outpatient visit

INTERVENTIONS:
Other: Virtual at Home Medication Reconciliation Visit(s) — Patients will have their medications reviewed by the TELE-TOC interventionalist, a member of the pharmacy team (anticipated)
  Other Names: Virtual At Home Medication Reconciliation
  Arms: TELE-TOC plus Usual Care
Behavioral: Virtual At Home Medication Education Visit(s) — Patients will be provided with inhaler education by the TELE-TOC interventionalist, a member of the pharmacy team (anticipated)
  Other Names: Virtual At Home Inhaler Education
  Arms: TELE-TOC plus Usual Care
Other: COPD advanced practice nurse Inpatient Consult — Patients will receive a COPD consult by an advanced practice nurse as part of standard of care
  Other Names: Inpatient consult
Other: Inpatient Medication Reconciliation — Patients will have their medications reviewed by member(s) of the clinical care team as part of standard of care
Other: Post-discharge nurse 48 hour phone follow-up call — Patients will receive a post-discharge nurse 48 hour phone follow-up call as part of standard of care
Other: Post-discharge follow-up advanced practice nurse outpatient visit — Patients will be scheduled for a 1-2 week post-discharge visit with the COPD advanced practice nurse as part of standard of care

SUMMARY:
Transitions of Care (TOC) between hospital, ambulatory, and home settings for high-risk, frequently hospitalized adults with chronic diseases, such as chronic obstructive pulmonary disease (COPD) are complex, costly, and vulnerable to safety threats and poor health outcomes. One potential solution to address this gap in care is the Transitional Care Model (TCM), which utilizes a patient-centered approach with in-home interventions; since in-person in-home visits are costly, using innovative telehealth, such as virtual visits via teleconferencing may be just as effective with greater feasibility, scalability, and sustainability, particularly in the post-COVID-19 era as has been seen the rapid expansion of these technologies. With a transdisciplinary team of experts from cognitive science, care transitions/handoffs, human factors engineering, design, implementation science, and health services research, the study team proposes to implement and evaluate via a randomized clinical trial the "TELE-TOC: Telehealth Education: Leveraging Electronic Transitions Of Care for COPD patients," intervention which includes a virtual visit, pharmacy-based, in-home intervention for COPD patients to improve medication use and patient outcomes among a population at high risk for readmission and medication safety events.

DETAILED DESCRIPTION:
Transitions of Care (TOC) for high-risk, frequently hospitalized adults with chronic diseases are complex, costly, and vulnerable to safety threats and poor health outcomes. Communication breakdowns, information lapses, and IT-induced unintended consequences can result in poor follow-up and medication non-adherence, both of which contribute to preventable readmissions or emergency room (ER) visits. The Transitional Care Model (TCM) aims to reduce such risks through a holistic, collaborative, patient-centered approach with in-home interventions. Prior to the coronavirus disease 2019 (COVID-19) pandemic, most in- home interventions relied on in-person visits, which can be cost-prohibitive and unsustainable. One potential sustainable and scalable solution is to use telehealth for in-home virtual visits; however, use of telehealth for post-discharge TOC interventions has not been routinely implemented. In the post-COVID-19 era, given the rapid expansion of telehealth, hospitals are well-positioned to initiate this virtual care. In-home virtual visits may be particularly promising for patients with chronic obstructive pulmonary disease (COPD), who are often hospitalized, have multiple comorbidities, and require intensive medication teaching due to rampant inhaler misuse. COPD affects more than 16 million US adults, many of whom are older, contribute ~$50 billion to healthcare costs annually, experience high rates of acute care revisits, often due to care coordination failures. For this reason, Medicare's Hospital Readmission Reduction Program (HRRP) aims to incentivize hospitals to implement TOC programs for increased quality and value of care for COPD patients. However, currently, such programs fall short of aligning with the full TCM. In-home interventions may be particularly salient for improving medication skills and outcomes for patients with COPD given rampant inhaler misuses, the effectiveness of in- hospital inhaler education, and evidence showing the need for inhaler education reinforcement post discharge. Thus, our trans-disciplinary team proposes to implement and evaluate "TELE-TOC: Telehealth Education: Leveraging Electronic Transitions Of Care for COPD patients," which seeks to integrate virtual, pharmacy-based, in-home visits for COPD patients within our hospital's existing COPD HRRP. The central hypotheses are that virtual visits with pharmacists will be feasible to implement and will result in improved medication use and outcomes among COPD patients at high risk for readmission. The investigator aims to iteratively design TELE-TOC using participatory study design and stakeholder input. The study team will then test the effectiveness of adding TELE-TOC virtual visits in a randomized controlled trial among COPD patients enrolled in the HRRP program. Lastly, the study team will develop a plan for a dissemination strategy and roadmap with national stakeholders to facilitate wide scale adoption of TELE-TOC nation wide.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Admitted to the hospital on a general inpatient ward with a COPD Exacerbation
* Enrolled/seen by our COPD Hospital Readmission Reduction Program

Exclusion Criteria:

* Patients younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Correct inhaler technique 30 days post discharge | 30 days post discharge
  Correct inhaler technique within 30 days post-discharge compared to baseline technique in hospital based on standardized checklists (<75% correct steps = misuse)
Reach of the TELE-TOC intervention | 1-2 weeks post discharge
  Proportion of patients receiving at home inhaler education within 1-2 weeks post discharge

SECONDARY OUTCOMES:
30 day revisits | 30 -days
  proportion of patients with any emergency department visit and/or re-hospitalization within 30 days of index admission
90 day revisits | 90 -days
  proportion of patients with any emergency department visit and/or re-hospitalization within 90 days of index admission
180 day revisits | 180 -days
  proportion of patients with any emergency department visit and/or re-hospitalization within 180 days of index admission
Medication errors | Within 30 days
  Proportion of patients with medication errors at TELE-TOC visit medication reconciliation
COPD Symptoms option 1 | Within 30 days
  Evaluation of COPD symptoms using COPD Assessment Test (CAT)
COPD Symptoms option 2 | Within 30 days
  Evaluation of COPD symptoms using the modified medical Research Council Scale (mmRC) [Scale = 0 to 4; 0 (better) = Breathlessness only on strenuous exercise; 4 (worse)= too breathless to leave the house or breathless when dressing or undressing]

CONTACTS AND LOCATIONS:
Overall Officials: Valerie G Press, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data, associated documentation, and study materials will be made available to other researchers following publication of the primary results. Data will be shared in accordance with institutional policies and data use agreements.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Naylor MD, Aiken LH, Kurtzman ET, Olds DM, Hirschman KB. The care span: The importance of transitional care in achieving health reform. Health Aff (Millwood). 2011 Apr;30(4):746-54. doi: 10.1377/hlthaff.2011.0041. PMID 21471497
- [Background] Locke ER, Thomas RM, Woo DM, Nguyen EHK, Tamanaha BK, Press VG, Reiber GE, Kaboli PJ, Fan VS. Using Video Telehealth to Facilitate Inhaler Training in Rural Patients with Obstructive Lung Disease. Telemed J E Health. 2019 Mar;25(3):230-236. doi: 10.1089/tmj.2017.0330. Epub 2018 Jul 17. PMID 30016216
- [Background] Thomas RM, Locke ER, Woo DM, Nguyen EHK, Press VG, Layouni TA, Trittschuh EH, Reiber GE, Fan VS. Inhaler Training Delivered by Internet-Based Home Videoconferencing Improves Technique and Quality of Life. Respir Care. 2017 Nov;62(11):1412-1422. doi: 10.4187/respcare.05445. Epub 2017 Jul 18. PMID 28720676
- [Background] Jencks SF, Williams MV, Coleman EA. Rehospitalizations among patients in the Medicare fee-for-service program. N Engl J Med. 2009 Apr 2;360(14):1418-28. doi: 10.1056/NEJMsa0803563. PMID 19339721
- [Background] Press VG, Au DH, Bourbeau J, Dransfield MT, Gershon AS, Krishnan JA, Mularski RA, Sciurba FC, Sullivan J, Feemster LC. Reducing Chronic Obstructive Pulmonary Disease Hospital Readmissions. An Official American Thoracic Society Workshop Report. Ann Am Thorac Soc. 2019 Feb;16(2):161-170. doi: 10.1513/AnnalsATS.201811-755WS. PMID 30707066
- [Derived] Ramadurai D, Lee CT, Traeger L, Pucci G, Jackson-Sagredo A, Shah S, Abraham J, Arora VM, Press VG. Telehealth Education Leveraging Electronic Transitions Of Care for COPD Patients (TELE-TOC): a study protocol for a type II hybrid effectiveness-implementation randomised, pragmatic clinical trial of a pharmacist-led intervention. BMJ Open. 2025 Nov 4;15(11):e105521. doi: 10.1136/bmjopen-2025-105521. PMID 41193196
- See also: Contextual Frameworks for Research on the Implementation of Complex System Interventions — https://www.ncbi.nlm.nih.gov/books/NBK196199
- See also: Centers for Medicare and Medicaid Services Hospital Readmission Reduction Program (HRRP) — https://www.cms.gov/medicare/medicare-fee-for-service-payment/acuteinpatientpps/readmissions-reduction-program